CLINICAL TRIAL: NCT01694160
Title: Consultant in Nephrology. MD., Ph.D.
Brief Title: Oral Paricalcitol in Renal Transplant Recipients for Reducing Albuminuria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Hallvard Holdaas, Consultant Nephrology, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/107 D; 2012-000429-32 (EudraCT Number)
Record Dates: First submitted 2012-09-23; First posted 2012-09-27 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Proteinuria
Keywords: kidney transplant patients; Albuminuria
MeSH Terms: conditions — Proteinuria; Albuminuria | interventions — paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paricalcitol (Experimental): Paricalcitol 2 ug/daily for 48 weeks
  Interventions: Drug: Paricalcitol
- no intervention (No Intervention)

INTERVENTIONS:
Drug: Paricalcitol — Zemplar (paricalcitol) 2ug daily, oral intake
  Arms: Paricalcitol

SUMMARY:
The main objective of this study is to examine if paricalcitol may reduce progression of graft fibrosis and proteinuria in kidney transplant patients. Cyclosporine and tacrolimus have a detrimental long-term effect by inducing graft fibrosis. About 50% of graft losses are related to interstitial fibrosis. Paricalcitol is a vitamin D receptor activator indicated for treatment of secondary hyperparathyroidism. Paricalcitol is known to exert an anti-inflammatory and antifibrotic and attenuate cyclosporine-induced fibrosis. Paricalcitol is also shown to be renoprotective by reducing proteinuria. No randomized controlled trials with paricalcitol are performed in renal transplant patients examining the effect on proteinuria and graft fibrosis.

DETAILED DESCRIPTION:
77 randomized, 37 paricalcitol, 40 no treatment

ELIGIBILITY:
Inclusion Criteria:

* kidney transplant patients

Exclusion Criteria:

* Previously transplanted

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in albumin/creatinine ratio from baseline to end of study. | 1 year
  Albumin will be measured in spot urine as albumin/creatinine ratio in mg/mmol. Assuming a type 1 error of 5% and at type II error of 20 %, with a clinically relevant difference in 3.5 mg/mmol from a baseline value of 15.0 + 10 mg/mmol the estimated number of patients in each arm should be 65, assuming a correlation between start and end value of 0.5.

CONTACTS AND LOCATIONS:
Overall Officials: Hallvard Holdaas, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Renal Section, Oslo University Hospital, Rikshospitalet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Yes

REFERENCES:
- [Derived] Pihlstrom HK, Ueland T, Michelsen AE, Aukrust P, Gatti F, Hammarstrom C, Kasprzycka M, Wang J, Haraldsen G, Mjoen G, Dahle DO, Midtvedt K, Eide IA, Hartmann A, Holdaas H. Exploring the potential effect of paricalcitol on markers of inflammation in de novo renal transplant recipients. PLoS One. 2020 Dec 16;15(12):e0243759. doi: 10.1371/journal.pone.0243759. eCollection 2020. PMID 33326471
- [Derived] Ussif A, Pihlstrom H, Pasch A, Holdaas H, Hartmann A, Smerud K, Asberg A. Paricalcitol supplementation during the first year after kidney transplantation does not affect calcification propensity score. BMC Nephrol. 2018 Aug 22;19(1):212. doi: 10.1186/s12882-018-1000-8. PMID 30134956